CLINICAL TRIAL: NCT00005960
Title: A Phase II Study of Doxorubicin and Cyclophosphamide With Sequential Docetaxel in Patients With Hormone-Refractory Prostate Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amgen (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067942; AMGEN-GCSF-980282; NCI-V00-1595
Record Dates: First submitted 2000-07-05; First posted 2004-06-08 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-01

CONDITIONS: Pain; Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; pain
MeSH Terms: conditions — Pain; Prostatic Neoplasms | interventions — Filgrastim; Cyclophosphamide; Docetaxel; Doxorubicin; Analgesia

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Procedure: pain therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the PSA response, duration of PSA response, disease free survival, median survival, and overall survival in patients with chemotherapy naive hormone refractory adenocarcinoma of the prostate treated with doxorubicin and cyclophosphamide with sequential docetaxel. II. Assess for any improvement in pain over time in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive doxorubicin IV over 3-5 minutes and cyclophosphamide IV on days 1, 22, 43, and 64, and docetaxel IV over 1 hour on days 85, 106, and 127 in the absence of disease progression or unacceptable toxicity. Patients receive filgrastim (G-CSF) subcutaneously daily beginning 24 hours after completion of chemotherapy infusions and continuing until blood counts recover. G-CSF must be discontinued at least 24 hours prior to starting subsequent chemotherapy infusions. Pain and analgesic use are assessed before study, every 3 weeks during study, after completion of study, and then at 3 months after completion of study. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter until death.

PROJECTED ACCRUAL: Approximately 42-105 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven adenocarcinoma of the prostate that is chemotherapy naive and refractory to hormonal therapy with combined androgen blockade No concurrent antiandrogen therapy withdrawal: Must continue antiandrogen therapy until completion of study OR Must discontinue flutamide at least 4 weeks before or bicalutamide at least 8 weeks before study enrollment, and must have disease progression off antiandrogen therapy, defined by serial increase in PSA (at least 2 measurements taken at least 2 weeks apart) or measurable tumor Concurrent LHRH antagonist allowed if no prior orchiectomy No minimum PSA level required Measurable or evaluable disease An increase in PSA or pain without measurable or evaluable disease does not constitute hormone refractory disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: SGOT and SGPT no greater than 2 times upper limit of normal Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF normal No impaired cardiac status (e.g., history of severe heart disease, cardiomyopathy, or congestive heart failure) Other: No active infection, defined by the following: Clinical syndrome consistent with a viral or bacterial infection (e.g., influenza, upper respiratory infection, or urinary tract infection) Fever with a clinical site of infection identified Microbiologically documented infection including, but not limited to, bacteremia or septicemia HIV negative No other malignancy within the past 5 years except surgically cured basal cell or squamous cell skin cancer No psychiatric, addictive, or other disorder that would preclude informed consent or compliance No hypersensitivity to E. coli derived proteins or drugs formulated with polysorbate 80 (e.g., human insulin)

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent WBC transfusions No other concurrent biologic therapy Chemotherapy: See Disease Characteristics No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: No other concurrent investigational agent No concurrent acetaminophen for fever prophylaxis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Debra Litwak, PharmD, Study Chair — Amgen
Locations (6):
- United States (6):
  - Wilshire Oncology Medical Group, Inc., Los Angeles, California
  - Geffen Cancer Center and Research Institute, Vero Beach, Florida
  - Arena Oncology Associates, Great Neck, New York
  - New York Medical College, Valhalla, New York
  - N.W. Carolina Oncology & Hematology, P.A., Hickory, North Carolina
  - Associates of Hematology/Oncology, Upland, Pennsylvania